CLINICAL TRIAL: NCT04075214
Title: Delivering Transcutaneous Auricular Neurostimulation (tAN) to Improve Symptoms Associated With Opioid Withdrawal
Brief Title: Transcutaneous Auricular Neurostimulation (tAN) for Symptoms of Opioid Withdrawal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spark Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SBM-OWP-02
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-07

CONDITIONS: Opioid-use Disorder; Opioid Withdrawal
Keywords: auricular neurostimulation; vagus nerve stimulation; transcutaneous; withdrawal symptoms
MeSH Terms: conditions — Opioid-Related Disorders; Substance Withdrawal Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- delayed-active tAN (Sham Comparator)
  Interventions: Device: transcutaneous auricular neurostimulation (tAN)
- active tAN (Experimental)
  Interventions: Device: transcutaneous auricular neurostimulation (tAN)

INTERVENTIONS:
Device: transcutaneous auricular neurostimulation (tAN) — Phoenix tAN system

SUMMARY:
Clinical performance data for transcutaneous auricular neurostimulation (tAN) as a method to aid in the reduction of symptoms associated with opioid withdrawal in order to support clinical substantial equivalence to a predicate device.

DETAILED DESCRIPTION:
Prior evidence has demonstrated that non-invasive neurostimulation can modulate specific brains regions associated with opioid use disorder and reduce opioid withdrawal symptoms. This is a double blind, randomized, controlled, multi-center study in which subjects will be randomized in a 1:1 ratio to one of two groups: 1) active transcutaneous auricular neurostimulation (tAN) or 2) delayed-active tAN to determine reduction of symptoms related to opioid withdrawal. Subjects in the active tAN group will receive tAN immediately whereas those in the delayed-active tAN will have their therapy turned on after a 30 minute delay (inactive period). All subjects will be informed of their group assignment at the conclusion of the randomized, double blind period (following initial 30 minutes of active or inactive therapy) and all will continue to receive active tAN throughout the five-day study. Each clinical site will have pre-determined and qualified clinical opiate withdrawal scale (COWS) accessor(s) that will be blind to the subjects group designation during the randomized, double blind period and will not be informed that all subjects receive active therapy throughout the remainder of the study. This will ensure a non-biased assessment of the COWS score and maintain single blinding throughout the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Current opioid dependence; prescriptive or non-prescriptive
2. COWS score is ≥ 13 or in the opinion of the investigator the subject is in moderate to severe withdrawal
3. 18-65 years of age
4. English Proficiency
5. Participants must be able to provide informed con-sent and function at an intellectual level sufficient for study requirements

Exclusion Criteria:

1. Current evidence of an uncontrolled and/or clinically significant medical condition
2. History of seizures or epilepsy
3. History of neurological diseases or traumatic brain injury
4. Participants using long-acting opioids such as methadone or buprenorphine for a period of five or more consecutive days prior to enrollment
5. Recent suicide attempt leading to current hospital admission or continued expressed suicidal ideation
6. Presence of devices, e.g. pace-makers, cochlear prosthesis, neuro-stimulators
7. Abnormal ear anatomy or ear infection present
8. Women of childbearing potential, not using adequate contraception as per investigator judgment or not willing to comply with contraception for the duration of the study
9. Females who are pregnant or lactating
10. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Clinical opiate withdrawal scale (COWS) score | 60 minutes
  Mean percent change in clinical opiate withdrawal scale (COWS) score from baseline to 60 minutes after start of active tAN therapy. The COWS is an 11-item scale with a score range between 0 and 48. Total score is the sum of all the items and a higher score indicates more severe withdrawal symptoms. Scores between 5 and 12 indicate mild withdrawal, scores between 13 and 24 indicate moderate withdrawal, scores between 25 and 36 indicate moderately severe withdrawal and scores greater than 36 indicate severe withdrawal. A COWS score reduction of 15% or greater for a given individual is considered clinically significant.

SECONDARY OUTCOMES:
Clinical opiate withdrawal scale (COWS) score | 30 minutes
  Comparison of mean percent change in COWS score in delayed active tAN versus active tAN groups at 30 minutes
Clinical opiate withdrawal scale (COWS) responder rate | 30 minutes
  Comparison of the proportion of participants with a clinically significant reduction in COWS score (defined as a 15% or greater reduction) in delayed-active tAN versus active tAN groups at 30 minutes
Clinical opiate withdrawal scale (COWS) score | 30 minutes
  Mean percent change in COWS score from baseline to 30 minutes after start of active tAN therapy
Clinical opiate withdrawal scale (COWS) score | 120 minutes
  Mean percent change in COWS score from baseline to 120 minutes after start of active tAN therapy
Clinical opiate withdrawal scale (COWS) score | Days 2-5
  Mean percent change in COWS score from baseline to Days 2 through 5 after start of active tAN therapy

OTHER OUTCOMES:
Heart rate variability measured by R to R interval | Days 2-5
  Mean change from baseline to Days 2-5 in heart rate variability measured by R to R interval
C-reactive protein (CRP) levels | Day 5
  Mean change in C-reactive protein (CRP) levels from baseline to Day 5
Cortisol levels | Day 5
  Mean change in cortisol levels from baseline to Day 5
Cytokine levels | Day 5
  Mean change in cytokine levels from baseline to Day 5
Patient Health Questionnaire (PHQ-9) | Day 5
  Mean change in depression symptoms measured by Patient Health Questionnaire (PHQ-9) total score from baseline to Day 5. The PHQ-9 is a nine-item depression scale based directly on the nine diagnostic criteria for major depressive disorder in the DSM-IV. Each of the nine items is rated on a 0 (not at all) to 3 (nearly every day) scale. A total score is calculated by summing the nine items. Scores range from 0 to 27 and higher scores indicate a higher degree of depression.
Post-Traumatic Stress Disorder (PTSD) Checklist for DSM-5 (PCL-5) | Day 5
  Mean change in PTSD symptoms measured by the PTSD Checklist for DSM-5 (PCL-5) total symptom severity score from baseline to Day 5. The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. Each of the 20 items is rated on a 0 (not at all) to 4 (extremely) scale. A total symptom severity score is calculated by summing the 20 items. Scores range from 0 and 80 and higher scores indicating a higher degree of PTSD symptomology. Evidence suggests that a10-20 point reduction in score represents a clinically significant change in PTSD symptoms.
World Health Organization Quality of Life - BREF (WHOQOL-BREF) | Day 5
  Mean change in WHOQOL-BREF domain scores (physical health, psychological health, social relationships, environment, and overall QoL/general health) from baseline to Day 5. The World Health Organization Quality of Life - BREF (WHOQOL-BREF) is a 26-item, self-report questionnaire which assesses 4 quality of life domains: physical health, psychological health, social relationships, and environment. In addition, there are 2 items that measure overall quality of life and general health. Subjects rate how much they have experienced each item in the preceding 2 weeks on a 5-point Likert scale ranging from 1 (not at all) to 5 (completely). Domain scores are scaled in a positive direction with higher scores denoting higher quality of life. Raw domain scores will be converted to a 0 to 100 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Navid Khodaparast, PhD, Study Director — Spark Biomedical, Inc.
Locations (1):
- Recovery Unplugged, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tirado CF, Washburn SN, Covalin A, Hedenberg C, Vanderpool H, Benner C, Powell DP, McWade MA, Khodaparast N. Delivering transcutaneous auricular neurostimulation (tAN) to improve symptoms associated with opioid withdrawal: results from a prospective clinical trial. Bioelectron Med. 2022 Aug 18;8(1):12. doi: 10.1186/s42234-022-00095-x. PMID 35978394